CLINICAL TRIAL: NCT02594150
Title: Single Center Randomized Pilot Study Of Colorectal Cancer Screening Outreach
Acronym: CRCSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 823388
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- usual care (No Intervention): Each FIT kit will include a tube in which to deposit the stool sample, directions on how to collect and mail the sample, a letter about colorectal cancer screening, a Labcorp requisition form, and a pre-paid return envelope.
- unconditional fixed incentive (Experimental): This arm will receive a FIT kit as described in the mailed FIT arm and will also receive a financial incentive in the form of a gift card and a note explaining that this gift card is a token of our appreciation for completing the kit.
  Interventions: Other: Financial Incentive
- conditional fixed incentive (Experimental): This arm will receive a FIT kit as described in the mailed FIT arm and will receive a note stating that they will receive a financial incentive in the form of a gift card if they return their completed FIT within two months of receiving the FIT kit.
  Interventions: Other: Financial Incentive
- conditional lottery incentive (Experimental): This arm will receive a FIT kit as described in the mailed FIT arm and will receive a note stating that they will be entered in a 1/10 chance lottery to receive a financial incentive in the form of a gift card if they return their completed FIT within two months of receiving the FIT kit.
  Interventions: Other: Financial Incentive

INTERVENTIONS:
Other: Financial Incentive — Financial incentives provide small immediate and tangible rewards that are aligned with the abstract long-term rewards of cancer prevention.
  Arms: conditional fixed incentive; conditional lottery incentive; unconditional fixed incentive

SUMMARY:
A four arm randomized pilot study to assess if the rate of completion of Fecal Immunochemical Test is increased by the addition of financial incentives.

DETAILED DESCRIPTION:
This is a single center 4-arm randomized pilot study to assess if the rate of completion of Fecal Immunochemical Test (FIT) is increased by the addition of financial incentives. Potentially eligible subjects will be identified via a data abstraction by Penn Data Store. We will conduct Electronic Medical Record (EMR) reviews on randomly select patients from the data abstraction using PennChart to confirm eligibility until 1,080 patients are identified. We will then randomize these 1,080 patients to one of four arms during the intervention phase.

* Arm 1: mailed FIT kit (usual care)
* Arm 2: mailed FIT kit + a gift card included in mailing (unconditional fixed incentive)
* Arm 3: mailed FIT kit + guarantee of receiving a gift card if kit is returned within two months (conditional fixed incentive)
* Arm 4: mailed FIT kit + entry in a 1/10 chance lottery to receive a gift card if kit is returned within two months (conditional lottery incentive) All 1,080 subjects will receive the mailed FIT kit. Subjects whose FIT results are not recorded in PennChart will receive a follow-up phone call via Interactive Voice Response (IVR) three weeks after the kit was mailed to the subject. Subjects whose FIT results are not recorded in PennChart will receive a follow-up mailed reminder six weeks after the kit was mailed to the subject. Subjects will receive follow-up regardless of the arm to which they are randomized.

A random sub-sample of 200 subjects will be called at least twelve weeks after the kit was mailed to the subject to complete a questionnaire. Verbal consent will be obtained from this sub-sample. This phone call will occur after the intervention and follow-up phases are completed. Analysis will occur after the sub-sample questionnaire phase is completed.

ELIGIBILITY:
Inclusion Criteria:

* Between 50 to 75 years old
* Has had at least two visits at Penn Family Care Within the past two years - Due for screening
* Asymptomatic for colorectal cancer (CRC)
* Zip code listed in PennChart as part of the subjects address is within the Philadelphia-Wilmington-Camden Metropolitan Statistical Area
* Have a primary care provider in Penn Family Care

Exclusion Criteria:

* Has had prior colonoscopy within 10 years, sigmoidoscopy within 5 years, and fecal occult blood test (FOBT)/FIT within twelve months of the chart review (We will exclude patients who self-report undergoing any of the above procedures)
* Has a history of CRC
* Has a history of other GI cancer
* Has history of confirmed Inflammatory Bowel Disease (IBD) (e.g. Crohn's disease, ulcerative colitis; Irritable bowel syndrome does not exclude patients)
* Has history of colitis other than Crohn's disease or ulcerative colitis
* Has had a colectomy
* Has a relative that has been diagnosed with CRC
* Has been diagnosed with Lynch Syndrome (i.e. HNPCC)
* Has been diagnosed with Familial Adenomatous Polyposis (FAP)
* Has anemia (iron-deficient or general/unspecified)
* Has history of lower GI bleeding
* Has metastatic (Stage IV) blood or solid tumor cancer
* Has end stage renal disease
* Has had congestive heart failure
* Has dementia
* Has cirrhosis or end stage liver disease
* Has any other condition that, in the opinion of the investigator, excludes the patient from participating in this study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 897 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Increase in return rate of completed FIT | 2 months
  An increase in return rate of completed FIT between intervention arms when compared to the control arm

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD MBA MSHP, Principal Investigator — University of Pennsylvania; Chyke Doubeni, MD MPH, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Derived] Mehta SJ, Pepe RS, Gabler NB, Kanneganti M, Reitz C, Saia C, Teel J, Asch DA, Volpp KG, Doubeni CA. Effect of Financial Incentives on Patient Use of Mailed Colorectal Cancer Screening Tests: A Randomized Clinical Trial. JAMA Netw Open. 2019 Mar 1;2(3):e191156. doi: 10.1001/jamanetworkopen.2019.1156. PMID 30901053